CLINICAL TRIAL: NCT05624216
Title: Radiofrequency and Targeted Pressure Energy for Cellulite Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-084_100
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Cellulite; Cellulitis; Cellulitis of Leg
MeSH Terms: conditions — Cellulite; Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- BTL-084 Treatment (Experimental): Radiofrequency and targeted pressure energy devices for the treatment of cellulite
  Interventions: Device: BTL-084

INTERVENTIONS:
Device: BTL-084 — Radiofrequency and targeted pressure energy devices for the treatment of cellulite
  Other Names: Emtone

SUMMARY:
This study will evaluate the clinical efficacy and safety of radiofrequency heating and targeted pressure energy for reduction in the appearance or cellulite. The study is a prospective multi-center open-label single-arm study. Subjects will be required to complete four (4) treatment visits and two to three follow-up visits - 1, 3 and 6 months after the last therapy visit. All of the study subjects will receive the treatment with the subject device.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and safety of radiofrequency heating and targeted pressure energy for reduction in the appearance or cellulite. The study is a prospective multi-center open-label single-arm study. Subjects will be required to complete four (4) treatment visits and two to three follow-up visits - 1, 3 and 6 months after the last therapy visit. All of the study subjects will receive the treatment with the subject device.

At the baseline visit subject's weight will be recorded, together with hip and thigh circumference. In addition, photographs of the treated area will be taken.

The treatment administration phase will consist of four (4) treatments, delivered in 2-4 weeks. The applicator will be applied over the treatment area.

At the last therapy visit, the subject's weight will be recorded, together with hip and thigh circumference. Photographs of the treated area will be taken. In addition, subjects will receive Subject Satisfaction Questionnaire and Therapy Comfort Questionnaire to fill in.

Safety measures will include documentation of adverse events (AE). Following each treatment administration and at all of the follow-up visits, subjects will be checked for immediate post-procedure adverse event assessment.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form
* Age ≥ 21 years
* Subject suffer from Grade 2 or Grade 3 cellulite as per Nürnberger-Muller Scale
* Subject did not experience weight change exceeding 2.5 kg (5 lb) in the preceding month
* BMI ≤ 33 kg/m2
* Women of childbearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote skin tightening and cellulite reduction during study participation
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without affecting significant change in either direction during study participation

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Autoimmune disease
* Diabetes
* Herpes Simplex
* Isotretinoin in the past 12 months
* Scleroderma
* Radiation therapy
* Burns in the treatment area
* Poor healing in the treatment area
* Metal implants
* Implantable pacemaker or automatic defibrillator / cardioverter
* Ablative / non-ablative cosmetic intervention (deep peeling) in the past 3 months
* Cancer and tumor diseases
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy / nursing or IVF procedure
* Acute neuralgia and neuropathy
* Blood disorders, risk of bleeding, bleeding tissues, peptic ulcers
* Eczema
* Rosacea
* Febrile conditions
* Kidney or liver failure
* Pronounced edemas, ascites, exudates
* Sensitivity disorders in the treatment area
* Varicose veins
* Local corticosteroid therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of cellulite severity change based on photographs before and after the study procedure according to the Cellulite Severity Scale | 6 months
  Three independent evaluators will evaluate photographs for a level of cellulite severity by assigning a score according to the Cellulite Severity Scale (CSS) validated by Hexsel et al. After follow-up visits are conducted, evaluators will be given a set of the coded photographs from each subject for an evaluation. The Cellulite Severity Scale evaluates five key morphological features of cellulite; number of depressions, depth of depressions, clinical appearance of evident raised lesions, presence of flaccidity and the grade of cellulite. Each item is graded from 0 to 3, allowing final classification of cellulite as mild, moderate and severe.
Photography evaluation according to the Global Aesthetic Improvement scale | 6 months
  Three independent evaluators will evaluate photographs for a level of appearance change by assigning a score according to the Global Aesthetic Improvement scale, where the lowest possible grade is (-1), worsened state and the highest is (3) very much improved.
Hip and Thigh Circumference Measure | 6 months
  Hip and thigh circumference measurements will be conducted at the baseline visit, after the last treatment and during all follow-up visits.

SECONDARY OUTCOMES:
Therapy Comfort | 6 months
  The 10-point scale will be used for evaluating the comfort during the study treatment. Subjects will be evaluating the comfort/discomfort on a scale from 1 ("No discomfort") to 10 ("Unbearable discomfort")
Subject Satisfaction | 6 months
  The 5-point Likert scale Satisfaction questionnaire will be used to evaluate the participant's satisfaction with the therapy outcome. The subjects will be answering questions with possible answers varying from "Strongly disagree" to "Strongly agree"

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Busso Cosmetic Dermatology, Coconut Grove, Florida, United States

IPD SHARING:
Plan to Share IPD: No